CLINICAL TRIAL: NCT00696982
Title: The Effect of Sitagliptin on Hypertension, Arterial Stiffness, Oxidative Stress and Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Shlomit Koren MD, Assaf-Harofeh Medical Center internal medicine A
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: shlomit9
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Diabetes Mellitus; Arterial Stiffness
Keywords: Arterial stiffness; Augmentation index; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): diabetic patients who are treated with metformin wiyh HBA1C>7% will get sitagliptin
  Interventions: Drug: sitagliptin
- B (Experimental): diabetic patients who are treated with metformin with HBA1C>7% will get glibenclamide
  Interventions: Drug: glibenclamide

INTERVENTIONS:
Drug: sitagliptin — sitagliptin 100 mg once daily for 3 months
  Arms: A
Drug: glibenclamide — glibenclamide 5 mg once a day titrated as neede up to 20 mg a day
  Arms: B

SUMMARY:
Recently a new category of antihyperglycemic therapy aiming to modulate the incretin system has emerged. These drugs induce insulin secretion without inducing hypoglycemia. The effect of the incretin modulators drugs on hypertension, arterial stiffness, inflammation and oxidative stress parameters have not been fully investigated yet.GLP-1 analogue has been suggested to have an effect on endothelium and the development of hypertension. Nystrom et al have demonstrated that GLP-1 improves endothelial dysfunction in a small group of type 2 diabetes subjects, with coronary heart disease. We hypothesize that DPP-4 inhibitor will have an effect on hypertension and arterial stiffness by effect on the NO pathway.The aim of this study is to investigate the effect of two insulin inducers drugs, sulfonyl urea and DPP-4 inhibitor on 24 hours blood pressure monitoring, arterial stiffness, oxidative stress and inflammation.

DETAILED DESCRIPTION:
Background:

Recently, a new category of hypoglycemic therapy has emerged, aimed to modulate the incretin system in diabetic patients. Compared to other drugs that induce insulin secretion, these agents do not cause hypoglycemia. However, until now the differential effects of incretin modulators and the classical insulin inducers on hypettension, arterial stiffness, inflammation and oxidative stress parameters have not been yet investigated.

Incretins The increase in plasma insulin levels following oral administration of glucose usually exceeds the levels observed after intravenous glucose administration. The phenomenon is defined as incretin effect and has been attributed to the intestinal hormones which are released after oral glucose administration. The two most important incretin hormones are glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide 1 (GLP-1).

Incretin effect is reduced in type-2 diabetic patients. After oral glucose administration, both GIP and GLP-1 are secreted and rapidly inactivated by an enzyme dipeptidyl peptidase 4 (DPP-4). Accordingly, the half-life of active GLP-1 is less than 2 min (2). Both GIP and GLP-1 stimulate insulin secretion in a glucose-dependent manner. Moreover, GLP-1 has also been shown to increase islet cell neogenesis and differentiation, as well as reduce apoptosis of β-cells in rodents. (3-5). Incretins also affect glucagon secretion. GIP stimulates glucagon production (6) ,whereas GLP-1 inhibits synthesis of the latter (7). Differential effects of the two peptides on glucagon secretion may prove responsible for normalization of blood glucose after intravenous injection of GLP-1 but not after administration of GIP or its derivatives [7, 8]. Therefore, GLP-1 is the only incretin that has been applied for treatment for diabetes.

In addition to its direct insulin/glucagons activities, GLP-1 has other extra-pancreatic effects:

* It inhibits gastric emptying and small bowel motility , the effects being dependent on nitric oxide (NO) (8).
* It induces satiety through a central nervous system mechanism (9).
* There is some data suggesting that GLP-1 infusion improves LV function .
* rGLP-1 infusion significantly attenuated the development of hypertension in Dahl Salt sensitive rats [11]. In patients with type 2 DM, exenatide treatment for 2 years also resulted in improvement of blood pressure [12]
* GLP-1 exerts direct beneficial effects on endothelium-dependent vasodilatation in healthy non-diabetic non-smoking normotensive subjects [13].
* In type 2 diabetic subjects with coronary heart disease, GLP-1 infusion significantly increased relative changes in brachial artery diameter (i.e. improved endothelial dysfunction) [14].

Since the main limitation of GLP-1 from the pharmacokinetic point of view is its rapid inactivation by DPP- 4, two strategies have been developed. One strategy is the development of GLP-1 receptor agonists (GLP-1 mimetics) which are resistant to DPP-4, such as exenatide (Byetta). The other approach is to prevent inactivation of GLP-1 by inhibiting the DPP-4 enzyme activity.

DPP-4 inhibitors Mice with a genetic deletion of DPP-4 have increased glucose tolerance following oral glucose administration in association with augmented insulin secretion. [15] DPP-4 inhibitor in animal studies was shown to augments the active GLP-1 concentration, increase insulin secretion and improve glucose tolerance. [16, 17] Previous rodent studies have found that GLP-1 and its analogues may increase beta cell mass by stimulating islet neogenesis and differentiation and inhibiting apoptosis.[3]. Similar effect can be produced by DPP-4 inhibition [18, 19].

Sitagliptin Sitagliptin is one of the two most studied DPP-4 inhibitors (the other one being vildagliptin). It is a competitive reversible inhibitor of the enzyme.[20] It is an orally active drug that can be absorbed rapidly and efficiently. Hepatic insufficiency does not seem to alter the pharmacokinetics of this drug, however, renal insufficiency increases circulating levels of sitagliptin. [21] Sitagliptin proved to be a well tolerated and safe drug, both for monotherapy and for combination therapy with metformin or thiazolidiediones. Thus far, no drug interactions have been observed with the DPP-4 inhibitors. However, recently post-marketing reports of anaphylaxis, angioedema, and rashes, including Stevens-Johnson syndrome, have emerged in sitagliptin treated patients. [22] The reported numbers of hypoglycemic events have been very low, as should be expected from the glucose- induced GLP-1 secretion/effect.

Sitagliptin has been shown to reduce HBA1C by 0.8%-1.1% , to decrease fasting plasma glucose and to increase beta cell function indices in type 2 diabetes patients, as a single therapy or in combination with metformin or thizolidinediones, as compared to placebo [23-27]. Sitagliptin and glipizide have similar effect on plasma glucose when administered in combination with metformin therapy. [28]

Arterial stiffness and endothelial dysfunction Augmentation of arterial blood pressure, reflecting the pulsatile component of blood pressure and thus arterial stiffness, is a well-known risk factor for cardiovascular disease outcome.[29-33] Augmentation index (AIx) measurement, a non-invasive way of appreciating the rate of arterial stiffness, has been shown to predict coronary artery disease (CAD) in whole population as well as in patients with type 2 diabetes [32, 34, 35]. Differential effects of the drugs on arterial stiffness may be, in part, responsible for the diversity of impacts of various antihypertensive drug/treatments on CAD.[33] The Conduit Artery Function Evaluation (CAFE) study, a sub-study to the Anglo-Scandinavian Cardiac Outcomes Trial (ASCOT), examined the impact of two different blood pressure lowering regimens, atenolol-thiazide based versus amlodipine-perindopril based therapy, on derived central aortic pressure values and on hemodynamics in 2199 patients.[33] Central pulse pressure was an independent risk factor for composite outcome of total cardiovascular events/procedures and the development of renal impairment. Similarly, statin drugs have been shown to exert additional beneficiary effects on AIx, the result entirely independent of their primary, cholesterol lowering, effect.[36]. Regarding type 2 diabetes, it has been previously demonstrated that increase in adiponectin levels, secondary to treatment with the insulin sensitizers pioglitazone or metformin, may decrease arterial stiffness.[37] . By analogy, incretins, in addition to stimulatory effects on insulin secretion, might have a positive impact on decreasing arterial stiffness in diabetic patients. Nystrom et al. have demonstrated that GLP-1 improves endothelial dysfunction in a small group of type 2 diabetes subjects with coronary heart disease [14]. However, the actual effect of DPP-4 on arterial stiffness has not yet been investigated.

According to the American diabetes association, treatment with biguanides should be started in case of diagnosis of type 2 diabetes .If the targeted glycemia level is not achieved, another medication should be added. In this respect, one cannot overemphasize the importance of discovering positive additional effects, if any, of the administered antidiabetic drugs on blood pressure, arterial stiffness, and oxidative stress and/or inflammation markers. The purpose of the proposed clinical trial is to compare the effects of two different types of insulin inducers, sulfonyl urea and incretin, on blood pressure, monitored within a 24h period, as well as on arterial stiffness parameters. In addition, assessment of blood markers for oxidative stress, as represented by 8-STAT-Isoprostane, oxidized LDL and [H202? carbonil groups?], as well as of markers for inflammation, as represented by TGF-ß, Il-1, Il-6, Il-4, Il-10 and highly sensitive CRP will be performed .

Methods The study has been designed as a prospective, randomized, single blind, cross-over trial. It will include 60 diabetic patients, aged 18 years or older, treated with metformin. Only patients with HbA1C levels within the range 7% - 11% will be enrolled in the study. All patients will submit written informed consent to participate in the experiment prior to their inclusion in the study.

The exclusion criteria will be as follows:

* CCT<30
* A history of treatment with incretins or sulfonylurea during the last 3 months
* Treatment with nitrates
* Uncontrolled heart failure
* Uncontrolled hypertension and/or any change in the hypertensive medications within one month prior starting the study
* No proven regular treatment with aspirin or statins within one month prior starting the study
* Any malignancy with life expectancy of less then 1 year
* pregnancy

Patients included in the study will be randomly assigned to one of the two experimental groups: Group A: to receive sitagliptin, 100 mg by a single dose daily, Group B: glibenclamide, 5 mg by a single dose daily. The latter dosage might be increased, if needed, to 5 mg twice a day. After 3 month, a one-week wash-out period during which no antidiabetic drugs (excluding metformin) will be administered, will be imposed on all patients .Following 1 week, a cross-over protocol will be applied: group A, earlier treated with sitagliptin, will now receive glibenclamid and, vice versa, group B will start the sitagliptin treatment.

The primary end results aimed to be obtained from this study are detection of arterial stiffness, defined as change in augmentation index measured by means of a non-invasive technique using the commercially available SphygmoCor System, and the results of the 24 hour blood pressure monitoring. The secondary end results would be oxidative stress parameters, as evaluated by oxidized LDL and Isoprostanes, and markers of inflammatory status, including measurements of pro-inflammatory interleukins and performance of highly sensitive CRP test.

All the patients enrolled in the study will be invited to the Research & Development Unit of Assaf-Harofeh for three visits: prior to starting the experiment, following 3 months and following 6 months. Their weight and abdominal circumference will be recorded; arterial stiffness will be measured; then, they will be connected to a blood pressure halter, recording their blood pressure for 24h. At each visit, 10ml periohera blood will be drawn for evaluation of HBA1C, complete blood count, serum electrolytes, albumin, blood lipids, fasting glucose 8F-STAT-Isoprostanes, oxidized LDL, nitric oxide, inflammatory interleukins and highly sensitive CRP (hsCRP). Any side effects of the drugs and any complaint on the event of hypoglycemia will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients
* aged 18 years or older
* treated with metformin
* Only patients with HbA1C levels within the range 7% - 11% will be enrolled in the study

Exclusion Criteria:

* CCT<30
* A history of treatment with incretins or sulfonylurea during the last 3 months
* Treatment with nitrates
* Uncontrolled heart failure
* Uncontrolled hypertension and/or any change in the hypertensive medications within one month prior starting the study
* No proven regular treatment with aspirin or statins within one month prior starting the study
* Any malignancy with life expectancy of less then 1 year
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
arterial stiffness, defined as change in augmentation index measured by means of a non-invasive technique using the commercially available SphygmoCor System, and the results of the 24 hour blood pressure monitoring | 6 months

SECONDARY OUTCOMES:
The secondary end results would be oxidative stress parameters, as evaluated by oxidized LDL and Isoprostanes, and markers of inflammatory status, including measurements of pro-inflammatory interleukins and performance of highly sensitive CRP test. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Koren, MD, Principal Investigator — Department of Internal Medicine A , Research & Development unit Assaf Harofeh Medical Center, Zerifin, affiliated to Sackler School of Medicine, Tel Aviv, Israel
Locations (1):
- Department of Internal Medicine A , Research & Development unit Assaf Harofeh Medical Center, Zerifin, affiliated to Sackler School of Medicine, Tel Aviv, Israel, Zrifin, Israel